CLINICAL TRIAL: NCT06678815
Title: How Can Volunteers in the NHS Be Best Supported?
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 347570; NIHR206121(08) (Other: NIHR (UK)); 347570 (Other: IRAS (UK))
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Those either working as, with, or treated by Community First Responders: Those either working as, with, or treated by Community First Responders
  Interventions: Other: Emergency response

INTERVENTIONS:
Other: Emergency response — Those delivering or receiving emergency care from a CFR.

SUMMARY:
This study aims to investigate the impact of volunteers in the English National Health Service (NHS) and increase the evidence base for supporting and developing volunteering to best help patients and services. The research will focus on one relatively established role: Community First Responders (CFR) supporting the ambulance service in English NHS Ambulance Trusts. We will take a mixed methods approach, combining qualitative and quantitative methods to learn more about the effectiveness and wider perceived value of the CFR role from the perspectives of CFRs themselves, other NHS staff and NHS patients who may interact with them.

Our primary Research Question is: How can we maximise the impact of the Community First Responder role? Secondary Research Questions focus on what we can learn from the Community First Responders to support volunteer roles more widely. In particular: How can policy makers improve the deployment of volunteers? How do staff perceive the support they receive from volunteers (including impact on their workload and morale)? How do patients perceive the support they receive from volunteers? How are volunteers impacting services? What opportunities are there for further developing the volunteer role? We will work with (up to five) Ambulance Trusts already involved in the National Ambulance Volunteering Dashboard to extract quantitative data from existing management systems. These data will focus on (1) number and demographic characteristics of CFRs; (2) aggregate CFR activity (incidents attended, first on scene, responses times, response outcomes) and (3) CFR incident data (including location, time, category and CFR attendance). From these Trusts we will select 2 for qualitative data collection consisting of documentary analysis and semi-structured interviews with CFRs, NHS staff and patients. This research aims to generate evidence to inform decisions on where policymakers can most efficiently focus future volunteer interventions and how the NHS can best support volunteers in the system.

DETAILED DESCRIPTION:
Purpose & research design

The study has a clear purpose - to learn more about the impacts that volunteers may have upon how NHS services function and how volunteers and volunteering can be supported. Whilst there is some existing research on the use of volunteers in the NHS, there are significant gaps in our knowledge - for instance about the effectiveness of volunteering in general - and the CFR role in particular, as well as the inter- and intra-organisational impacts of volunteering and the CFR role. For instance, do patients welcome and value the work of CFRs? Likewise, do NHS staff integrate well with CFRs, or not?

The mixed method research design enables the research team to collect data on both the impacts that the CFR role has on NHS services whilst exploring the perceptions of CFRs themselves, the patients they serve and the NHS colleagues with whom they interact.

The multi-site research design enables the research team to compare findings from different geographical settings thereby enabling both particularisation and transferability.

Motivation and relevance

The invitation to conduct the research comes from the Department for Health and Social Care (DHSC). This reflects the policy salience of the work. It is strongly supported by the Association of Ambulance Chief Executives (AACE). For both the DHSC and AACE, the findings of the research will be of high value in relation to lessons for wider developments of volunteering in the NHS as well as refinement of the CFR role.

Recruitment & Selection

Recruitment decisions are led by AACE stakeholders. Pragmatism guides many of these decisions. It is important that the (Ambulance Trust) sites that are recruited are not only willing to take part but also able to provide the quantitative data of interest in a timely and efficient manner. 5 sites have been identified as both willing and able to provide these data and will be invited to take part based on the existing organisational knowledge of the AACE.

From within these 5 sites, we will purposively identify 2 sites for in depth qualitative data collection. We do not foresee any significant ethical, legal or managerial issues in relation to the collection, analysis and dissemination of the qualitative data that this study will generate.

In 2023 the AACE developed a National Ambulance Volunteering Dashboard (NAVD). This was designed to highlight the range of individuals who support ambulance trusts, the activities in which they participate, and the patients they help via clinical and non-clinical volunteering opportunities.

The quantitative element of this project will aim to build on this work to help the engaged trusts to identify and standardise their data relating to CFRs. This data is likely to be held on varying systems and using different categorisation and data linkages. Given limited resources in each trust we will need to work to identify which data can be accessed and extracted without disproportionate additional burden to the trusts. This may mean that the resulting data has elements missing and it is highly likely that trusts will vary in their capacity to provide data. We will minimise this risk by only reporting descriptive statistics from the trusts with transparent reporting on data gaps. The project can be used as a baseline with which the trusts can work to improve this data quality.

Where possible the data on CFRs will be combined with existing statutory collections for ambulance dispatch data relating to response times, categories, conveyance rates and other information. All data relating to CFRs will need to be anonymised within the trust and data suppression used to ensure that any data shared with the project has no risk of disclosure.

The qualitative work will consist of approximately 15 semi-structured interviews in each of the 2 qualitative sites (30 in total), with key informants (likely to include several CFRs with different levels of experience and career trajectories; NHS staff - Ambulance service strategic and operational managers, NHS ambulance service paramedics, ambulance service call handlers; Hospital Emergency Department staff - both clinical and managerial) and service users. These interviews will mostly take place virtually via Microsoft Teams.

We will request local policy documents produced by NHS Ambulance and NHS hospital Trusts that outline the roles and responsibilities of CFRs to triangulate the interview and focus group findings alongside publicly available national and regional documents.

Interviews

To recruit interview participants into the qualitative part of the study, we will draw on the support of the volunteer managers at each of our selected sites. These individuals are best placed to help the research team to identify and help approach service users, CFRs and NHS informants. The volunteer managers will reach out to potential informants and inform the potential informants about the research. If potential informants are happy to take part, then their email addresses will be shared with the research team. Potentially interested informants will then receive an individual email from a member of the researcher team with a participant information sheet inviting them to take part in the research project. A date and time for the online interview will be agreed between the informant and the researcher. Before the interview, the informant will be sent a consent form to complete. In the online meeting, the researcher will go through the information sheet and consent form with the informant and enable them to ask any questions they may have. Once consent is granted, the recording function will be enabled interview will be recorded. The interviews will most likely last about 60 minutes.

Each interview recording will be given an anonymised reference number. An audio file will be made of each interview and saved to the King's College London One Drive in a protected folder. Each anonymised audio file will be securely transferred for transcription by a professional transcriber. Following transcription, a word document will be securely shared with the research team - identifiable only by an anonymised reference number. This file will be uploaded into a securely located qualitative research software platform to enable the researchers to code and analyse the data further.

Documents

Any confidential documents that are shared with the research team such as protocols, strategy documents etc. will be treated in a similar way to interview transcripts - i.e., they will be given an anonymised identification code and uploaded into a qualitative research software platform for analysis alongside any publicly available documentation. The qualitative analysis will not include any documents will patient identifiable data.

Risks, burdens and benefits

Overall, there is a risk that these inquiries pose political risks to the trusts, if they are construed as trusts being reliant on volunteers to keep response times down, or using volunteers as a substitute for paid staff. It will be important that the narrative put around these data is careful to emphasise that volunteers add value rather than replace paid staff. In relation to the qualitative research specifically, there are no risks for those taking part in interviews or focus groups as all information will be fully anonymised. The only burden is that of participants' time. There are likely to be few direct personal benefits for individuals through taking part. However, there may be wider benefits for NHS patients, clinicians, managers and policy makers through the knowledge generated in this project through greater understanding of volunteering in the NHS.

Confidentiality

We will follow University and NHS best-practice Principles through each stage of this proposed research project as outlined above.

Conflicts of Interest

We do not foresee any conflicts of interest in the proposed research.

ELIGIBILITY:
Inclusion Criteria:

* working as/with or treated by CFR

Exclusion Criteria:

* not working as/with or treated by CFR

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those working as/with or treated by CFR
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Descriptive data on CFR demographics and activities | 2025
  Descriptive statistics on CFRs

SECONDARY OUTCOMES:
Qualitative data on CFR role/NHS volunteering more broadly | 2025
  Interview data

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.kcl.ac.uk/hscwru